CLINICAL TRIAL: NCT05743127
Title: 3D-Printed Versus Laboratory-Fabricated Hyrax Expanders: A Randomized Controlled Clinical Trial
Brief Title: 3D-Printed Versus Laboratory-Fabricated Hyrax Expanders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ildeu Andrade Jr. (Other)
Collaborators: American Association of Orthodontics Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Ildeu Andrade Jr., Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24070148
Record Dates: First submitted 2023-01-10; First posted 2023-02-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Expansion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group Conventional Expander (Experimental): Conventional Laboratory Fabricated Hyrax Expander
  Interventions: Device: Conventional Laboratory Fabricated Hyrax Expander
- Group 3-D Printed Expander (Experimental): 3D-Printed Hyrax Expander
  Interventions: Device: 3D-Printed Hyrax Expander

INTERVENTIONS:
Device: 3D-Printed Hyrax Expander — This is a type of maxillary expander that is designed on a computer and printed in metal using 3D printers and is used to expand the upper jaw.
  Arms: Group 3-D Printed Expander
Device: Conventional Laboratory Fabricated Hyrax Expander — This is a type of maxillary expander that is made by hand in an orthodontic laboratory and is used to expand the upper jaw.
  Arms: Group Conventional Expander

SUMMARY:
Maxillary expanders are orthodontic appliances that are commonly used to expand the upper jaw. The purpose of this study will be to compare the effects produced by two different maxillary expanders in children 8-13 years old. The first type of expander is made by hand in an orthodontic laboratory, and the second type of expander is designed on a computer and printed using 3D printers. Both expanders are already used in the MUSC Orthodontics Clinic. The purpose of this study is to see if the 3D printed expander is as effective as the traditional expander made by hand in the laboratory, with more comfort to the patient. Patients participating in the study will be randomly assigned to one of two groups: group A will be treated with a laboratory-made maxillary expander, and group B with a 3D-Printed maxillary expander. Information will be collected on the participants' standard clinical follow-up visits including photos, x-rays, and dental photo scans over the course of 6 months to see how the expander is working. In addition, as part of the research study, the participant will be asked to complete online questionnaires with assistance from parents or guardians about his/her quality of life and perception of possible pain and discomfort at different time points. The potential benefits of this study include the use of 3D technology to improve the quality of the orthodontic treatment, with more comfort to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary anterior and/or posterior transverse deficiency with or without crossbite
* Age of 8-13 years
* Children whose parents/guardians are willing to consent to the child participating in the study
* Children ages 12-13 who are willing to assent to participating in the study
* Children who are orthodontic patients at the Medical University of South Carolina Department of Orthodontics or University of Pittsburgh School of Dental Medicine
* Subjects and parents/guardians who have access to an electronic device with internet connection

Exclusion Criteria:

* Patients with previous or ongoing orthodontic treatment
* Patients whose parents have a strong preference as to which expander is used
* Patients with a history of temporomandibular disorders
* Presence of congenitally missing teeth
* Traumatic loss of maxillary incisors
* Patients with craniofacial syndromes, or cleft lip and/or palate

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Dimension of the Anterior Midpalatal Suture Opening | 2 weeks
  The dimension of the anterior midpalatal suture opening between the maxillary halves will be measured digitally in millimeters on the occlusal radiograph using a calibrated ruler.

SECONDARY OUTCOMES:
Change in Interincisal Diastema Width | 2 weeks
  The change in interincisal diastema width will be measured in millimeters on the post-expansion (T1) digital models between the maxillary central incisors using OrthoAnalyzer 3D software.
Change in Maxillary Molar Inclination | 2 weeks
  Using measurement tools in OrthoAnalyzer 3D software and the T0 digital models, the inter-molar inclination of the maxillary permanent first molars will be evaluated. The inclination of the T1 maxillary permanent first molars will be measured in a like-manner as the T0 digital models. The intermolar inclination measurement at T1 will be subtracted from the intermolar inclination measurement at T0 to record any presumably positive increase in molar inclination.
Change in Maxillary Arch Widths | 2 weeks
  The measurements of the maxillary dental arch widths will be performed on the pre-expansion (T0) and post-expansion (T1) digital models using the OrthoAnalyzer software. The intercanine, interpremolar or first deciduous molar, and intermolar widths will be measured in millimeters. The widths at T0 will be subtracted from the widths at T1 to record any positive increase in arch widths.
Pain Perception assessed by Visual Analog Scale | 2 weeks
  Using an online questionnaire, patients will be asked about the highest pain level they will have experienced at different time points using the visual analog scale (VAS). The higher the value in the VAS scale, the more severe the pain.
Pain Perception assessed by Wong-Baker FACES Scale | 2 weeks
  Using an online questionnaire, patients will be asked about the highest pain level they will have experienced at different time points using the Wong-Baker FACES Scale. The more upset the face in the Wong-Baker FACES Scale, the more severe the pain.
Oral Health Related Quality of Life (functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicap) assessed by OHIP-14 | 2 weeks
  Using an online questionnaire, patients will be asked about his/her quality of life at different time points using the short version of the Oral Health Impact Profile (OHIP-14). The OHIP-14 has 14 questions distributed across seven domains: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The scores for each domain and the total score will be evaluated. A higher score indicates a more negative perception of the individual with respect his/her quality of life. The lowest score is 0, which indicates a more positive perception of the individual with respect his/her quality of life. The highest score is 4, which indicates a more negative perception of the individual with respect his/her quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ildeu Andrade, DDS, MS, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh - School of Dental Medicine, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No